CLINICAL TRIAL: NCT06731582
Title: Targeting Metabolic Insufficiency (TAMING) Glaucoma Study : a 2-year Multi-centre, Double-masked, Randomised, Placebo-controlled Trial of Nicotinamide (Vitamin B3) Supplementation in Glaucoma
Brief Title: Nicotinamide Supplementation in Glaucoma
Acronym: TAMING
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Singapore Eye Research Institute (Other)
Collaborators: National University Hospital, Singapore (Other); Singapore National Eye Centre (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-2039; OFLCG21Jun-0014 (Other Grant/Funding Number: National Medical Research Council (NMRC))
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Glaucoma
Keywords: nicotinamide; vitamin B3; NAM
MeSH Terms: conditions — Glaucoma | interventions — Niacinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nicotinamide (Experimental): 1.5 grams/day (2 tablets of 750 mg each)
  Interventions: Dietary Supplement: Nicotinamide Tablet
- Placebo (Placebo Comparator): 2 tablets
  Interventions: Dietary Supplement: Nicotinamide Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide Tablet — 1.5 grams/day
  Arms: Nicotinamide
Dietary Supplement: Nicotinamide Placebo — 2 tablets
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if nicotinamide (NAM, vitamin B3) supplementation can delay glaucoma progression 30% above that achieved with conventional glaucoma treatment using topical medication. The main questions it aims to answer are:

Can NAM supplementation improve the visual function of patients with glaucoma measured by visual field perimetry?

Researchers will compare NAM to a placebo (a look-alike substance that contains no drug) to see if NAM works as an adjuvant in glaucoma treatment.

Participants will:

* Take NAM or a placebo every day for 2 years
* Visit the clinic once every 3-4 months for checkups and tests

DETAILED DESCRIPTION:
520 subjects with glaucoma will be enrolled (260 per study arm) from Singapore National Eye Centre and National University Hospital Eye Clinic.

The TAMING Glaucoma Study is designed as a phase 3, randomised, placebo-controlled, double-masked, superiority trial with two parallel groups and a primary endpoint of change in visual field progression over two-three years.

Participants who are currently on NAM will be asked to stop taking the tablets for a month prior to screening visit.

The study duration and your follow-up will be approximately 2-3 years. Recruitment: All participants will be sent an e-consent form via email or provided in hard copy for them to read. Participants will be allowed to ask questions and be given as much time as they require to consider whether they would like to participate. It will be made clear that it will not influence their clinical care in any way whether they agree to participate or not or choose to withdraw from the study at any given time. Written informed consent will be sought from participants prior to screening. Participants will be recruited from public and private ophthalmology clinics at the SNEC and NUH ophthalmology outpatient clinics.Research staff will screen medical records/medical history of patients attending glaucoma clinics to identify potential participants. A study team member will approach eligible patients to explain the study in detail either in person.

Screening visit: At screening, a participant's ophthalmic history will be taken to determine whether they are eligible for the study based on the ophthalmic inclusion and exclusion criteria.

Randomisation: Randomisation will be performed as block randomisation, stratified by glaucoma sub-type and trial site, with a 1:1 allocation.

After baseline testing, participants will be allocated to NAM or placebo in a ratio 1:1 utilising block randomisation stratified by glaucoma subtype and trial site. One or both eligible eyes will be enrolled. Statistical corrections will be used for bilaterally in the final analysis.Web-based randomisation will be conducted through REDCap. Research staff involved in data collection or assessing outcomes, statisticians and participants will remain masked to treatment allocation. A unique code will be allocated to each participant rather than a fixed code for each treatment group such that the unblinding of one individual will not affect the study group as a whole. Participants in the treatment group will take NAM (1.5 g/day - 2 tablets with food) for the remainder of the study.

Blinding: After baseline testing, participants will be allocated to NAM or placebo in a ratio 1:1 utilising block randomisation stratified by glaucoma subtype and trial site. Both eyes will be enrolled. Research staff involved in data collection or assessing outcomes, statisticians and participants will remain masked to treatment allocation. The period of supplementation for both the treatment and placebo group would be for 24 months.

EMERGENCY UNBLINDING: To maintain the overall quality and legitimacy of the clinical trial, code breaks should occur only in exceptional circumstances when knowledge of the actual treatment is absolutely essential for further management of the patient. The Principal Investigator should be made aware of such circumstances.The Investigator is encouraged to maintain the blind wherever possible. The Investigator must report all code breaks (with reason) as they occur on their electronic CRF on REDCap. As unblinding may not necessarily be a reason for study drug discontinuation, the actual allocation should not be disclosed to the participant or other members of the research team.

Test procedures: Refraction, Central cornea thickness, best corrected visual acuity, Blood pressure measurement, Urine Pregnancy test, slit lamp biomicroscopy, intra ocularpressure measurement, visual field testing, Fundus imaging, optical coherence tomography, electroretinography (optional), blood sampling for liver tests - Alanine transaminase / aspartate aminotransferase (ALT/AST) and genetics testing , Patient reported outcome measures (PROMs) Questionaire, Health Economic Evaluation (optional).

Discontinuation / withdrawal: the investigator may withdraw a subject from the study treatment if he is in violation of the protocol, experiences a serious or intolerable adverse event, develops symtopms/ conditions listed in the exclusion criteria during the study, wishes to withdraw from treatment. The investigator will also withdraw allsubjects from the study treatment if the study is terminated. Individuals who discontinue the study treatment will be encouraged to continue in the study and complete the evaluations.They are free to withdraw from the study at any time upon their request or the request of their legally acceptable representative. When a subject withdraws from the study, the reasons for withdrawal will be recorded by the investigator. Whenever possible, all subjects who withdraw from the study prematurely will continue to undergo scheduled visits for study assessments (follow-up). Subjects who fail to return for study assessments will be contacted by the research team in an attempt to have them comply with the protocol, by two documented phone calls and one email. Subjects who withdraw will not be replaced and sample size calculation accounts for 15% attrition. If voluntary withdrawal occurs, the subject will be asked to continue scheduled evaluations, complete an end of study evaluation, and be given appropriate care under medical supervision until the symptoms of any adverse event resolve or the subject's condition becomes stable.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ³ 21 years, with definitive, treated POAG, PACG including normal tension glaucoma, PDG, PXFG in one or both eyes.

  * Best-corrected visual acuity equal or better than 6/18
  * Reproducible visual field defect due to glaucoma (3 contiguous points at less than 5%) and severity of visual field loss, MD between -2 and -18 dB. This range includes people with moderate disease which optimises detection of progression.
  * Patients must have at least two prior 24-2 VF tests which meet <16% FP and <21% fixation loss.
  * Previous selective laser trabeculoplasty is acceptable (IOP-lowering laser treatment) if ³ 3 months prior or filtering surgery >6 months previously.
  * Normal liver function tests.
  * Those taking NAM already will undergo a 1-month washout period bef

Exclusion Criteria:

* Patients with active liver disease or end stage renal failure.

  * Active use of allopurinol, carbamazepine, or primidone.
  * Visually significant cataracts (example, likely to require surgery within 2 years).
  * Cataract surgery in the last 3 months or glaucoma filtration surgery in last 6 months.
  * Conditions that may cause non-glaucomatous visual field defect (for example, severe ptosis, cerebrovascular accident, prior panretinal photocoagulation, and other retinal or central nervous system diseases).
  * Not able to complete study (for example, concurrent severe systemic disease).
  * History of cancer in the last 5 years.
  * Unable to give consent.
  * Inability to tolerate or take nicotinamide and/or pyruvate.
  * Women of Child Bearing Potential, pregnancy or lactation.
  * History of Hypotension
  * Blood Pressure measurement of less than 90/60(

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Mean Deviation (MD) | 2 years
  ≥ 30% reduction in visual field mean deviation progression measured over 2 years compared to current IOP-lowering treatments alone.

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore, Central Singapore
  - Singapore Eye Research Institute, Singapore, Central Singapore

IPD SHARING:
Plan to Share IPD: Undecided